CLINICAL TRIAL: NCT01246349
Title: Motivational Interviewing as an Intervention to Increase Adolescent Self-Efficacy and Promote Weight Loss
Brief Title: Motivational Interviewing for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Staff Endocrinologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000017625
Record Dates: First submitted 2010-11-11; First posted 2010-11-23 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Childhood Obesity
Keywords: Motivational Interviewing; Child and Adolescent Self-Efficacy; Health Behaviours
MeSH Terms: conditions — Pediatric Obesity | interventions — Motivational Interviewing; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing Group (Experimental): For the Motivational Interviewing (MI) treatment group, a clinical psychology doctoral student trained in Motivational Interviewing administered six individual motivational interviewing treatment sessions, each 30 minutes in length.
  Interventions: Behavioral: Motivational Interviewing (Treatment Group)
- Control Group (Active Comparator): The comparison group received six social skills training sessions instead of Motivational Interviewing (MI).
  Interventions: Behavioral: Social Skills Training (Control Group)

INTERVENTIONS:
Behavioral: Motivational Interviewing (Treatment Group) — Motivational interviewing (MI) can be defined as a client-centered, directive method of therapy for enhancing intrinsic motivation to change by exploring and resolving ambivalence (Miller and Rollnick, 2002). MI manifests through specific strategies, such as reflective listening, summarization, shared decision making, and agenda setting.
  Arms: Motivational Interviewing Group
Behavioral: Social Skills Training (Control Group) — Within the social skills training framework, advice is given to clients and sessions are focused on assigning goals for clients to work towards without specific regard for their readiness to change. The intervention is aimed at finding appropriate ways to navigate typical social situations (e.g., how to negotiate with parents).
  Arms: Control Group

SUMMARY:
The investigators studied the effect of motivational interviewing (MI) on self-efficacy, health behaviors, and health outcomes in overweight children and adolescents (ages ranging from 10 to 18 years).

DETAILED DESCRIPTION:
One empirically supported intervention with a large evidence base for improving adult outcomes in behavioral health-related disorders is Motivational Interviewing (MI). MI is strongly rooted in the client-centered therapy of Rogers (1951). Its relational stance emphasizes the importance of understanding the client's internal frame of reference and displaying unconditional positive regard for the client. Motivational interviewing can thus be defined as a client-centered, directive method of therapy for enhancing intrinsic motivation to change by exploring and resolving ambivalence. MI manifests through specific strategies, such as reflective listening, summarization, shared decision making, and agenda setting.

Adolescent participants exposed to motivational interviewing in conjunction with usual care (diet and exercise program) are expected to endorse greater self-efficacy, report increased engagement in healthy behaviors, demonstrate a decrease in body weight and report improved psychological outcomes. While motivational interviewing has been shown to increase adults' motivation to make healthy behavior changes, few adolescent studies have demonstrated this effect.

ELIGIBILITY:
Inclusion Criteria:

* Obese youth (with Body Mass Index (BMI) ≥ to 85th percentile for age and gender (as classified by the Center for Disease Control))
* ages 10-18 years
* attending a local obesity clinic ("Healthy Weights" clinic)

Time of entry into the weight-loss program was controlled for; however, both new and current participants had the option to participate in the study.

Exclusion Criteria:

* taking medication whose side effects may influence weight gain or weight loss
* did not speak English
* demonstrated a developmental delay
* reported being pregnant and/or reported having an eating disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overweight and obese youth (BMI ≥ 85th %ile for age and gender) were eligible to participate and were recruited directly by the primary investigators from the Toronto East General Hospital's Healthy Lifestyles program, comprised of children and adolescents ages 10-18 years who are seeking diet and exercise treatment for their obesity.
Pre-assignment Details: Individuals were excluded if they: 1) were taking medication whose side effects may influence weight gain or weight loss, 2) did not speak English, 3) had a known developmental delay, and 4) reported being pregnant and/or having an active eating disorder.
Groups:
- Control Group: The control group received social skills training in place of motivational interviewing, conducted over 6 months by an interventionist not trained in MI to avoid cross-contamination.
  The social skills interventionist used a standardized treatment manual, developed and validated for children and adolescents. The social skills interventionist offered advice (as opposed to eliciting ideas from the client, as is the case with MI) and clients were assigned goals to work on without specific regard for the clients' readiness to change. Sessions were based around finding appropriate ways to navigate typical social situations (for example, how to negotiate with parents, how to manage emotions or how to make friends).
- Treatment/Experimental Group: The Treatment group received Motivational Interviewing (MI). MI is a client-centered, directive method of therapy for enhancing intrinsic motivation to change by exploring and resolving ambivalence (Miller and Rollnick, 2002). MI manifests through specific strategies, such as reflective listening, summarization, shared decision making, and agenda setting.
  A clinical psychology doctoral student trained in MI administered the intervention over the course of 6 months to participants assigned to the treatment group. The MI intervention comprised six individual MI treatment sessions, each approximately 30 minutes in length.
Period: Overall Study
Arm/Group | Control Group | Treatment/Experimental Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group (Motivational Interviewing): The treatment group received Motivational Interviewing (MI), which is a client-centered, directive method of therapy aimed at enhancing a client's intrinsic motivation to change by exploring and resolving ambivalence.
  MI utilizes strategies to guide the patient, as opposed to offering advice or focusing on accomplishing specific goals. For example, using reflective listening and shared decision making are common within the MI approach.
  Six individual MI sessions, approximately 30 minutes in length each, were provided by a trained clinical psychology doctoral student.
- Control (Social Skills Training): The control group received social skills training in place of Motivational Interviewing (MI). The social skills training was provided by a therapist who was not trained in MI to avoid cross-contamination.
  The social skills training provided was a standardized and manualized treatment, developed and validated for children and adolescents. As part of this training, the interventionist offered advice and clients were assigned specific tasks to work on. No consideration of clients' readiness to change was made in this group.
- Total: Total of all reporting groups
Arm/Group | Treatment Group (Motivational Interviewing) | Control (Social Skills Training) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.8) | 13.7 (1.7) | 13.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Weight Efficacy Life-style Questionnaire
Description: A self-efficacy instrument, the Weight Efficacy Life-style Questionnaire (WEL; Clark, Abrams, Niaura, Eaton, & Rossi, 1991) was used to measure participants' beliefs about and confidence in their own ability to make a behavior change, specifically their ability to lose weight.
  The questionnaire yields a total score, with higher scores indicating higher levels of health-related self-efficacy, as well as 5 situational sub-scores (negative emotions, availability, social pressure, physical discomfort, and positive activities). Individuals rate statements on a 10-point scale ranging from 0 (not confident) to 9 (very confident).
  The WEL is made up of 20 items (4 items per sub-scale) which are summed to obtain a total score, with the lowest total score possible being 0 and the highest 180. Only the total WEL score was used in the study's analyses.
  The difference in self-efficacy (WEL) change between treatment and control groups from baseline to a 6 month follow-up was examined.
Time Frame: Baseline, 6 month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Motivational Interviewing Group: The Treatment group received Motivational Interviewing (MI). MI is a client-centered, directive method of therapy for enhancing intrinsic motivation to change by exploring and resolving ambivalence (Miller and Rollnick, 2002). MI manifests through specific strategies, such as reflective listening, summarization, shared decision making, and agenda setting.
  A clinical psychology doctoral student trained in MI administered the intervention over the course of 6 months to participants assigned to the treatment group. The MI intervention comprised six individual MI treatment sessions, each approximately 30 minutes in length.
Arm/Group | Control Group | Motivational Interviewing Group
Number analyzed (Participants) | 20 | 20
scores on a scale
  Baseline WEL | 120.70 (29.32) | 128.80 (27.24)
  Follow-up WEL | 139.88 (19.88) | 136.40 (26.77)
Statistical Analysis 1: Comparison: Control Group vs Motivational Interviewing Group; Published results comprise baseline and follow-up means and standard deviations for both the MI and control group (reported above), as well as the absolute attributable effect of intervention (i.e., the difference in self-efficacy [WEL] change between the treatment and control groups from baseline to a 6 month follow-up); Test type: Superiority or Other; p = 0.24, Regression, Linear; Mean Difference (Final Values) = 8.616, 95% CI 2-sided [-5.871 to 23.103], Standard Error of Mean 7.373

2. Secondary Outcome: Physiological Outcomes: BMI
Description: The study used a Body Mass Index (BMI) percentile for age as the main indicator of weight-loss. Height and weight was measured by the pediatrician at the treatment site and BMI as well as BMI percentile for age was determined with the use of an age appropriate growth curve chart.
Time Frame: Baseline, 6 month follow-up
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Control Group | Motivational Interviewing Group
Number analyzed (Participants) | 20 | 20
z-score
  Baseline BMI | 2.64 (0.73) | 2.51 (0.47)
  Follow-up BMI | 2.41 (0.78) | 2.46 (0.47)
Statistical Analysis 1: Comparison: Control Group vs Motivational Interviewing Group; Results published comprise baseline and follow-up BMI z-score means and standard deviations for both the MI and control groups (reported above), as well as the attributable effect of intervention (i.e., the difference in BMI change between the treatment and control groups from baseline to a 6-month follow-up); Test type: Superiority or Other; p = 0.56, Regression, Linear

3. Secondary Outcome: Physiological Outcomes: Waist Circumference
Description: Measurements of waist circumference, an indirect measure of central adiposity (or fatness), were also obtained.
Time Frame: Baseline, 6 month follow-up
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control Group | Motivational Interviewing Group
Number analyzed (Participants) | 20 | 20
cm
  Baseline Waist Circumference | 95.7 (11.4) | 92.8 (6.6)
  Follow-up Waist Circumference | 93.6 (10.9) | 94.35 (7.5)
Statistical Analysis 1: Comparison: Control Group vs Motivational Interviewing Group; Results published comprise baseline and follow-up means and standard deviations for both the MI and control group (reported above), as well as the attributable effect of intervention (i.e., the difference in waist circumference change between the treatment and control groups from baseline to a 6-month follow-up); Test type: Superiority or Other; p = 0.09, Regression, Linear

4. Secondary Outcome: Psychological Well-being
Description: Rosenberg Self-Esteem scale, Pediatric Quality of Life Inventory (PEDS QL), Child depression inventory, Adolescent coping (A-COPE)
Time Frame: Change over time from Baseline to 6 months (measured monthly) with a 12 months reassessment
Reporting Status: Not Posted

5. Primary Outcome: Child Dietary Self-Efficacy Scale
Description: A second self-efficacy scale, the Child Dietary Self-Efficacy Scale (CDSS; Parcel et al., 1995) was used to measure participants' confidence in their ability to choose lower fat, lower sodium foods.
  The questionnaire is made up of 20 likert items with 3 response options, including "not sure", "a little sure", and "very sure". Each item asks the participant to indicate how sure he/she is that they would make a healthy choice, for example, "How sure are you that you could eat cereal instead of a donut?" Individual items are scored -1, 0, or 1 and subsequently summed for a total score, with the lowest possible score a -20 and the highest a 20, whereby higher scores signify higher dietary self efficacy.
Time Frame: Baseline, 6 month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Motivational Interviewing Group
Number analyzed (Participants) | 20 | 20
scores on a scale
  Baseline CDSS | 9.35 (3.28) | 9.42 (4.53)
  Follow-up CDSS | 8.59 (3.26) | 8.55 (4.50)
Statistical Analysis 1: Comparison: Control Group vs Motivational Interviewing Group; Based on previous research , baseline CDSS means were expected between 5 - 6.5 with a SD of 3 - 4. It was hypothesized that an attributable effect of 1.5 would be detected. Published results comprise baseline and follow-up means and standard deviations for both the MI and control group (reported above), as well as the absolute attributable effect of intervention (i.e., the difference in self-efficacy [CDSS] change between the treatment and control groups from baseline to a 6 month follow-up); Test type: Superiority or Other; p = 0.88, Regression, Linear; Mean Difference (Final Values) = 0.183, 95% CI 2-sided [-2.301 to 2.668], Standard Error of Mean 1.265

ADVERSE EVENTS:
Arm/Group | Control Group | Motivational Interviewing Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No